CLINICAL TRIAL: NCT05667116
Title: An Observational Study to Assess the Real-world Effectiveness of EVUSHELD™ (Tixagevimab/Cilgavimab) as Pre-exposure Prophylaxis Against COVID-19 Among EVUSHELD-eligible Populations Receiving Care at UPMC in the United States
Brief Title: eVusheld Assessment reaL wORld Effectiveness at UPMC
Acronym: VALOR-C19 UPMC
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: D8850R00001
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: SARS-CoV-2, COVID-19
Keywords: EVUSHELD, AZD7442, SARS-CoV-2, COVID-19, Immunocompromise
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- EVUSHELD arm: 3,000 Individuals given EVUSHELD for pre-exposure prophylaxis
  Interventions: Drug: EVUSHELD
- Concurrent Control arm: 3,000 individuals eligible for EVUSHELD pre-exposure prophylaxis but did not receive Evusheld

INTERVENTIONS:
Drug: EVUSHELD — EVUSHELD (AZD 7442, Tixagévimab/Cilgavimab)
  Groups: EVUSHELD arm

SUMMARY:
An AstraZeneca-sponsored observational, electronic healthcare record (EHR)-embedded retrospective cohort study to assess the real-world effectiveness of EVUSHELD against SARS-CoV-2 infection, COVID-19-related hospitalization, and other COVID-19 related outcomes in the total EUA-eligible patient population in the University of Pittsburgh Medical Center (UPMC) Health System.

DETAILED DESCRIPTION:
This a Phase IV observational, secondary data study to assess the effectiveness of Evusheld in preventing COVID-19 infection and severe outcomes using the electronic medical records from the nationwide integrated health system.

The study is designed as an AstraZeneca-sponsored observational, electronic healthcare record (EHR)-embedded retrospective cohort study to assess the real-world effectiveness of EVUSHELD against SARS-CoV-2 infection, COVID-19-related hospitalization, and other COVID-19 related outcomes in the total EUA-eligible patient population in UPMC health system

ELIGIBILITY:
Inclusion Criteria:

1. Receipt of EVUSHELD under the FDA EUA for EVUSHELD
2. Eligibility for assess Evusheld use under the EUA. -

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All EVUSHELD EUA-eligible patient population in the UMPC health system.
Sampling Method: Non-Probability Sample
Enrollment: 4232 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
COVID-19 hospitalisation | 6 months
  To assess the effectiveness of EVUSHELD as PrEP against COVID-19 hospitalisation
All-cause mortality | 6 months
  To assess the effectiveness of EVUSHELD as PrEP against all-cause mortality

SECONDARY OUTCOMES:
SARS-CoV-2 infection | 6 & 12 months
  To assess the effectiveness of EVUSHELD as PrEP against documented SARS-CoV-2 infection
Medically attended COVID-19 | 6 & 12 months
  To assess the effectiveness of EVUSHELD as PrEP against medically attended COVID-19
Medically attended acute COVID-19 | 6 & 12 months
  To assess the effectiveness of EVUSHELD as PrEP against medically attended acute COVID-19
COVID-19 hospitalisation | 12 months
  To assess the effectiveness of EVUSHELD as PrEP against COVID-19 hospitalisation
COVID-19 intensive care unit (ICU) admission | 6 & 12 months
  To assess the effectiveness of EVUSHELD as PrEP against COVID-19 intensive care unit (ICU) admission

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Yealy, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Research Site, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted_CSR Synopsis_D8850R00001 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850R00001&attachmentIdentifier=82468668-cfb2-446d-a99d-46cded0732e6&fileName=Redacted_CSR_Synopsis_D8850R00001.pdf&versionIdentifier=